CLINICAL TRIAL: NCT01874821
Title: Adhesive Capsulitis and Dynamic Splinting: a Randomized, Controlled Trial
Brief Title: Adhesive Capsulitis and Dynamic Splinting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unrelated to trial
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010.005; SHD (Other: Dynasplint)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Adhesive Capsulitis
Keywords: Frozen Shoulder; Adhesive Capsulitis; ROM; Dynasplint
MeSH Terms: conditions — Bursitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynasplint (Experimental): Along with standard manual physical therapy, patients will have a stretching device (Dynasplint) used in rehabilitation to regain ROM in stiff joints. Patients will use this device 20-30 minutes 2 times per day at home.
  Interventions: Device: Dynasplint; Other: Standard of Care
- Control (Other): Patient's in the Physical Therapy Group will have the standard manual treatments during their usual physical therapy visits with no additional intervention
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Dynasplint — Dynamic splinting utilizes the protocols of Low-Load Prolonged Stretch (LLPS) with calibrated adjustable tension to increase Total End Range Time (TERT)to reduce contracture. The Dynasplint or "Experimental" group will add this therapy to their standard of care regimen
  Other Names: Shoulder
  Arms: Dynasplint
Other: Standard of Care — The current Standard of Care for treating this condition includes corticosteroid injections and physical therapy.

SUMMARY:
The purpose of this study is to examine the efficacy of dynamic splinting in reducing contracture following diagnosis of adhesive capsulitis.

DETAILED DESCRIPTION:
This randomized controlled trial will explore the efficacy of dynamic splinting in conjunction with the current standard of care as compared to standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 25% reduction in maximal external rotation plus greater than 25% reduction in at least one other plane of motion (elevation or abduction), as compared to the asymptomatic shoulder, measure supine with humerus abducted to 90º
* Duration from onset less than 12 months.
* Pain that is worsened by moving the arm in that direction

Exclusion Criteria:

* Any previous shoulder surgery.
* Brachial plexus injuries
* Neurologically mediated pain and fibromatosis-like contracture
* Concomitant neurologic complaints or abnormalities
* Glenohumeral impingement or mechanical blockage
* Oncological process affecting the shoulder
* Previous total mastectomy
* Glenohumeral arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 6 months
  The primary measures are full arc ROM and changes in the Disabilities of the Arm Shoulder Hand pain survey (DASH).

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

REFERENCES:
- [Background] Baums MH, Spahn G, Nozaki M, Steckel H, Schultz W, Klinger HM. Functional outcome and general health status in patients after arthroscopic release in adhesive capsulitis. Knee Surg Sports Traumatol Arthrosc. 2007 May;15(5):638-44. doi: 10.1007/s00167-006-0203-x. Epub 2006 Oct 10. PMID 17031613
- [Background] Castellarin G, Ricci M, Vedovi E, Vecchini E, Sembenini P, Marangon A, Vangelista A. Manipulation and arthroscopy under general anesthesia and early rehabilitative treatment for frozen shoulders. Arch Phys Med Rehabil. 2004 Aug;85(8):1236-40. doi: 10.1016/j.apmr.2003.12.032. PMID 15295746
- [Background] Farrell CM, Sperling JW, Cofield RH. Manipulation for frozen shoulder: long-term results. J Shoulder Elbow Surg. 2005 Sep-Oct;14(5):480-4. doi: 10.1016/j.jse.2005.02.012. PMID 16194738
- [Background] Hsu AT, Hedman T, Chang JH, Vo C, Ho L, Ho S, Chang GL. Changes in abduction and rotation range of motion in response to simulated dorsal and ventral translational mobilization of the glenohumeral joint. Phys Ther. 2002 Jun;82(6):544-56. PMID 12036396
- [Background] Rundquist PJ, Anderson DD, Guanche CA, Ludewig PM. Shoulder kinematics in subjects with frozen shoulder. Arch Phys Med Rehabil. 2003 Oct;84(10):1473-9. doi: 10.1016/s0003-9993(03)00359-9. PMID 14586914
- [Background] Vermeulen HM, Rozing PM, Obermann WR, le Cessie S, Vliet Vlieland TP. Comparison of high-grade and low-grade mobilization techniques in the management of adhesive capsulitis of the shoulder: randomized controlled trial. Phys Ther. 2006 Mar;86(3):355-68. PMID 16506872